CLINICAL TRIAL: NCT01088854
Title: Acute Effect of Continuous Positive Airway Pressure on Left Ventricular Diastolic Function and Exercise Tolerance in Compensated Heart Failure
Brief Title: Acute Effect of Continuous Positive Airway Pressure in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marjory Bussoni, mester, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: upeclin/HC/FMB-Unesp-30
Record Dates: First submitted 2009-10-16; First posted 2010-03-17 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2010-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- positive airway pressure (Experimental)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — unique session of 30-minute of continuous airway positive pressure

SUMMARY:
Acute effects of CPAP on diastolic function in patients with compensated heart failure (CHF) are unknown. The investigators hypothesized that acutely CPAP improves diastolic function, which is associated with increases exercise tolerance.

Objective: To evaluate the acute effects of CPAP on functional capacity and diastolic indices of patients with CHF. This is a randomized trial including 44 patients with compensated heart failure (functional classes II or III, NYHA). Patients will be allocated in CPAP(CPAP with 10cmH2O) or simulated CPAP (null pressure) after computed randomization, in a 1:1 ratio. All subjects shall complete a 6-minute walk test (6MWT) before and after CPAP (30 minutes; 10 cm H2O pressure). Doppler-echocardiogram will be performed before and at the end of CPAP. Wilcoxon or paired t tests were used to compare results, with significance level at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* functional class II or III (NYHA)heart failure
* agreement to participate in the study
* absence of acute exacerbation of dyspnea
* intact upper airway

Exclusion Criteria:

* valvular heart disease
* chest pain or unstable angina
* acute myocardial infarction in the prior month
* uncontrolled hypertension
* atrial fibrillation or other arrhythmias
* acute infection
* orthopedic limitations
* intolerance to CPAP mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
improvement of isovolumetric relaxation time | 30 minutes
  Doppler-derived isovolumetric time will be measured before and after intervention (CPAP). A decreasing in isovolumetric time after CPAP will be interpretated as an improvement in myocardial relaxation

SECONDARY OUTCOMES:
walk distance in the walk-test-six-minute (WT6M) | 30 minutes
  subjects will be tested before and after procedure (CPAP). An increasing distance after procedure will be interpretated as improved tolerance to exercise

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz B Matsubara, MD, Principal Investigator — Full Professor Botucatu Medical School; UNESP
Locations (1):
- UPECLIN - Botucatu Medical School, Botucatu, São Paulo, Brazil

REFERENCES:
- [Background] Bradley TD, Logan AG, Kimoff RJ, Series F, Morrison D, Ferguson K, Belenkie I, Pfeifer M, Fleetham J, Hanly P, Smilovitch M, Tomlinson G, Floras JS; CANPAP Investigators. Continuous positive airway pressure for central sleep apnea and heart failure. N Engl J Med. 2005 Nov 10;353(19):2025-33. doi: 10.1056/NEJMoa051001. PMID 16282177
- [Derived] Bussoni MF, Guirado GN, Matsubara LS, Roscani MG, Polegato BF, Minamoto ST, Bazan SG, Matsubara BB. Diastolic function and functional capacity after a single session of continuous positive airway pressure in patients with compensated heart failure. Clinics (Sao Paulo). 2014;69(5):354-9. doi: 10.6061/clinics/2014(05)010. PMID 24838902